CLINICAL TRIAL: NCT04236193
Title: Ultrasound and Immunological Findings in Patients With Shoulder Injury Related to Vaccine Administration (SIRVA)
Acronym: SIRVA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christoph Berger, PI Translational Immunology, University Hospital, Basel, Switzerland
Other Study IDs: SIRVA
Record Dates: First submitted 2019-11-15; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Shoulder Injury Related to Vaccine Administration; Erosion, Localized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SIRVA: Subjects with shoulder pain >7 days after vaccination
  Interventions: Diagnostic Test: Ultrasound Shoulder and Immunological Phenotyping by FACS
- Controls: Subjects from a prospective influenza vaccine study
  Interventions: Diagnostic Test: Ultrasound Shoulder and Immunological Phenotyping by FACS

INTERVENTIONS:
Diagnostic Test: Ultrasound Shoulder and Immunological Phenotyping by FACS — Cross-sectional Ultrasound exam of the affected shoulder. Peripheral blood measurements of the T and B cell subsets. Anti-Influenza Antibody measurements

SUMMARY:
Accidental vaccine injection into adjunct shoulder structures can cause tissue damage, termed Shoulder injury related to vaccine administration (SIRVA). The immunopathological mechanisms and consequences of SIRVA are unknown.

The study assesses the clinical and immunological consequences of an influenza vaccine if accidentally administered in periarticular space.

ELIGIBILITY:
Inclusion Criteria:

* participation at a local vaccination campaign
* Shoulder pain >3 days after vaccination

Exclusion Criteria:

* no vaccine received
* preexisting shoulder pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects receiving the Influenza vaccine at a local vaccination campaign in Basel, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pathological Findings in Ultrasound | Ultrasound of the shoulder is performed at Baseline/Inclusion
  Cross-sectional assessment and description of pathological ultrasound findings in subjects with shoulder pain after influenza vaccination

SECONDARY OUTCOMES:
Increased Vaccine response | Baseline and 12 months
  Antibodies against Influenza, Plasmablasts and T follicular helper cell increase

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Berger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Data on flowcytometry based immunophenotyping